CLINICAL TRIAL: NCT03709706
Title: A Phase 1b/2a Pilot Study to Evaluate the Safety and Tolerability of Autologous T-Cells Expressing Enhanced TCRs (T Cell Receptors) Specific for NY-ESO-1/LAGE-1a (GSK3377794) Alone, or in Combination With Pembrolizumab in HLA-A2+ Participants With NY-ESO-1- or LAGE-1a-Positive Advanced or Recurrent Non-Small Cell Lung Cancer
Brief Title: Pilot Immunotherapy Study With Letetresgene Autoleucel (Lete-cel, GSK3377794)T-cells in New York Esophageal Squamous Cell Carcinoma-1 (NY-ESO-1)/ LAGE-1a-positive Advanced Non-small Cell Lung Cancer (NSCLC) Either Alone or in Combination With Pembrolizumab
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated for reasons pertaining to feasibility
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 208471
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Neoplasms
Keywords: GSK3377794; Pembrolizumab; T Cell Receptors; Adoptive T-cell therapy; Non-Small Cell Lung Cancer; Immuno-oncology; NY-ESO-1; LAGE-1a; Leukapheresis; Letetresgene autoleucel
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Participants will receive GSK3377794, either as monotherapy or in combination with pembrolizumab.
Masking Description: This will be an open-label study. Hence, there will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: lete-cel monotherapy (Experimental): In Arm A, participants with NSCLC (lacking actionable genetic aberrations) will receive lete-cel monotherapy. Participants who subsequently progress by Week 25 will be offered pembrolizumab.
  Interventions: Drug: Lete-cel; Drug: Pembrolizumab
- Arm B: lete-cel plus pembrolizumab (Experimental): In Arm B, participants with NSCLC (lacking actionable genetic aberrations) will receive lete-cel followed by pembrolizumab.
  Interventions: Drug: Lete-cel; Drug: Pembrolizumab
- Arm C: lete-cel plus pembrolizumab (Experimental): In Arm C, participants with NSCLC (with actionable genetic aberrations) will receive lete-cel followed by pembrolizumab.
  Interventions: Drug: Lete-cel; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lete-cel — lete-cel will be administered to eligible participants.
Drug: Pembrolizumab — Pembrolizumab will be administered to eligible participants.

SUMMARY:
This trial will evaluate safety and tolerability of letetresgene autoleucel (GSK3377794) with or without pembrolizumab in participants with non-small cell lung cancer.

DETAILED DESCRIPTION:
New York esophageal squamous cell carcinoma-1 (NY-ESO-1) and LAGE-1a antigens are tumor-associated proteins that have been found in several tumor types. Clinical trials using adoptively transferred T- cells directed against NY-ESO-1/LAGE-1a have shown objective responses. Letetresgene autoleucel (GSK3377794) is the first generation of NY-ESO-1 specific T-cell receptor (TCR) engineered T-cells. This is a multi-arm, open-label study of letetresgene autoleucel (lete-cel, GSK3377794) in Human Leukocyte Antigen (HLA)-A*02:01, HLA-A*02:05 and/or HLA-A*02:06 positive adults whose tumors express NY-ESO-1 and/or LAGE-1a. This study will enroll participants who have unresectable Stage IIIb or Stage IV NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years on the day of signing informed consent.
* Histologically or cytologically diagnosed unresectable Stage IIIb or Stage IV NSCLC.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Participant is positive for any of the following alleles: human leukocyte antigen (HLA)-A*02:01, HLA-A*02:05, and a) or HLA-A*02:06 by a validated test.
* Participant's tumor meets the pre-defined threshold for expression of NY-ESO-1 and/or LAGE-1a.
* Adequate organ function and blood cell counts, as defined in the protocol.
* Predicted life expectancy that is >=24 weeks from leukapheresis.
* Left ventricular ejection fraction >=45%.
* Prior therapies prior to lymphodepletion: a) All participants with NSCLC lacking actionable genetic aberrations, per National Comprehensive Cancer Network (NCCN) guidelines (Arms A and B), need to have received at least one line of programmed death protein 1/programmed death protein 1 ligand (PD-1/PD-L1) checkpoint blockade therapy. For participants in the metastatic setting, PD-1/PD-L1 checkpoint blockade therapy must have been received either alone, in combination or sequentially with platinum-containing chemotherapy. OR b) All participants with NSCLC with actionable genetic aberrations, per NCCN guidelines (Arm C only), should have received appropriate targeted therapy following NCCN or equivalent country-level guidelines.
* Disease progression at time of treatment, as defined in the protocol.
* Measurable disease at time of treatment per response evaluation criteria in solid tumors (RECIST) version 1.1 as assessed by local site investigator/radiology.

Exclusion Criteria:

* Prior treatment: Previous treatment with genetically engineered NY-ESO-1-specific T-cells. Previous NY-ESO-1 vaccine or NY-ESO-1 targeting antibody. Prior gene therapy using an integrating vector.
* Prior allogeneic/autologous bone marrow or solid organ transplantation.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide, fludarabine, dimethylsulfoxide (DMSO) or other agents used in the study.
* Severe hypersensitivity (>= Grade 3) to pembrolizumab and/or any of its excipients.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* History of chronic or recurrent (within the last year prior to enrollment) severe autoimmune or active immune-mediated disease requiring steroids or other immunosuppressive treatments.
* Uncontrolled intercurrent illness.
* Participant has active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), Epstein Barr virus (EBV), cytomegalovirus (CMV), syphilis, or human T lymphotropic virus (HTLV), as defined in protocol.
* Known psychiatric or substance abuse disorders.
* Symptomatic or untreated central nervous system (CNS) metastases.
* Radiotherapy that involves the lung (Percentage of normal lung receiving at least 20 Gray [Gy] during radiotherapy [V20] exceeding 30% lung volume or mean heart dose >20 Gy) within 3 months or radiotherapy (including but not limited to palliative radiotherapy) to lung/mediastinum with V20 less than 30% lung volume and with mean heart dose <=20 Gy within 4 weeks (+/- 3 days).
* Radiotherapy of >=50 Gy to a significant volume of the pelvis, long bones or spine, or a cumulative dose of radiation that, in the investigator's opinion would predispose participants to prolonged cytopenia after lymphodepletion.
* All of the participant's measurable lesions have been irradiated within 3 months before lymphodepletion.
* Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (20):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Netherlands (4):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study that evaluated the safety and tolerability of autologous T-cells expressing enhanced T-cell receptors (TCRs) that were specific for New York esophageal squamous cell carcinoma (NY-ESO)-1 and/or Cancer testis antigen 2 (LAGE-1a) (GSK3377794, Lete-cel) in participants with Advanced or Recurrent Non-Small Cell Lung Cancer who had Human Leukocyte Antigen (HLA)-A02:01, HLA-A02:05, and/or HLA-A*02:06.
Pre-assignment Details: A total of 34 participants were enrolled in this study, out of which 13 received Lete-cel infusion. The study was terminated due to reasons pertaining to feasibility As a result of the early termination, no participants were assigned to Arm B, and thus no analysis of Arm B was performed.
Groups:
- Arm A: Lete-cel Monotherapy: Eligible participants underwent leukapheresis to manufacture autologous T cells bearing T- cell receptors (TCR) specific for NY-ESO-1/LAGE-1a. Lymphodepleting chemotherapy was administered, consisting of cyclophosphamide at a dose of 900 mg/m^2/day on day -7 through day -5 and fludarabine at a dose of 30 mg/m^2/day on day -8 through day -5. On day 1, participants received a single infusion of Lete-cel. Participants who had disease progression within 25 weeks of Lete-cel infusion were offered therapy with Pembrolizumab following benefit-risk evaluation. Pembrolizumab 200 mg was administered every three weeks (Q3W) for up to 35 cycles (up to Week 106) or until subsequent disease progression or intolerable toxicity. Pembrolizumab therapy was not allowed if disease progression occurred post 25 weeks of Lete-cel infusion.
- Arm C: Lete-cel + Pembrolizumab: Eligible participants underwent leukapheresis to manufacture autologous T cells bearing T-cell receptors (TCR) specific for NY-ESO-1 /LAGE-1a. Lymphodepleting chemotherapy was administered, consisting of cyclophosphamide at a dose of 900 mg/m^2/day on day -7 through day -5 and fludarabine at a dose of 30 mg/m^2/day on day -8 through day -5. On day 1, participants received a single infusion of Lete-cel followed by pembrolizumab 200 mg starting on Day 22 (Week 4 Day 1). Pembrolizumab was administered every three weeks (Q3W) for up to 35 cycles (up to Week 106) or until disease progression, whichever occurred first.
Period: Overall Study
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Started | 20 | 14
Intent-to-Treat (ITT) Population (Intent-to-Treat population includes all participants who started the leukapheresis procedure.) | 20 | 14
Modified - Intent to Treat Population (Includes all participants in ITT population who received Lete-cel infusion.) | 7 | 6
No Treatment (Participants who underwent leukapheresis but did not go on to receive lymphodepletion chemotherapy or Lete-cell infusion.) | 13 | 8
Completed (Participants who received Lete-cel infusion and were followed-up in this study until death or for 15 years after infusion, or until transfer to a separate long-term follow-up (LTFU) study and participants who completed the treatment but did not transfer to LTFU study because Protocol amendment 06 was not in place to allow the transfer, are considered to have completed the study.) | 3 (Three participants died after Lete-cel infusion.) | 3 (One participant was transferred to the long-term follow-up study, NCT03391778 (208750). Another participant died after Lete-cel infusion. A third participant completed the treatment but did not transfer to the LTFU study because the protocol amendment 06 was not in place to allow the transfer.)
Not Completed | 17 | 11
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 14 | 8
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death Prior to Lete-cel Infusion | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab | Total
Number analyzed (Participants) | 20 | 14 | 34
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 62.1 (8.90) | 59.4 (10.25) | 61.0 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 5 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  White | 19 | 12 | 31
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. AEs which start or worsen on or after T-cell infusion are defined as treatment-emergent.
Time Frame: Up to approximately 10 months
Population: Modified Intent-to-Treat (mITT) population included all participants who received Lete-cel infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 7 | 6
Participants
  AEs | 7 | 6
  SAEs | 5 | 3

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events of Special Interest (AESI)
Description: AESI included cytokine release syndrome (CRS), pneumonitis/pneumonia, graft vs host disease (GvHD), guillain barre syndrome (GBS) or acute inflammatory demyelinating polyneuropathy (AIDP), pancytopenia/aplastic anemia (including analysis of all hematopoietic cytopenias), immune effector cell-associated neurotoxicity syndrome (ICANS) and treatment-related inflammatory response at tumor site. AEs which start or worsen on or after T-cell infusion are defined as treatment-emergent.
Time Frame: Up to approximately 10 months
Population: Modified Intent to Treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 7 | 6
Participants | 6 | 6

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events and Serious Adverse Events Based on Maximum Severity Grades
Description: An AE is any untoward medical occurrence in a clinical investigation, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. AEs which start or worsen on or after T-cell infusion are defined as TE. Severity was reported during study and was assigned a grade according to the National Institutes of Health National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE). SAEs are subset of AEs. AEs and SAEs severity graded on a 5-point scale as: 1 = mild, 2 = moderate discomfort, 3 = severe, 4 = life-threatening and 5 = death due to AE.
Time Frame: Up to approximately 10 months
Population: Modified intent-to-treat (mITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 7 | 6
Participants
  AEs, Grade 2 | 1 | 0
  AEs, Grade 3 | 1 | 3
  AEs, Grade 4 | 5 | 2
  AEs, Grade 5 | 0 | 1
  SAEs, Grade 3 | 4 | 2
  SAEs, Grade 4 | 1 | 0
  SAEs, Grade 5 | 0 | 1

4. Primary Outcome: Number of Participants With AEs Leading to Dose Delays
Description: An AE is any untoward medical occurrence in a clinical investigation, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with AEs leading to dose delays were summarized.
Time Frame: Up to approximately 10 months
Population: Modified intent-to-treat (mITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 7 | 6
Participants | 1 | 1

5. Primary Outcome: Overall Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Investigator Assessment
Description: Overall response rate (ORR) defined as the percentage of participants with a complete response (CR) or partial response (PR) via investigator assessment per RECIST (Response Evaluation Criteria in Solid Tumors Criteria) v1.1 relative to the total number of participants in the analysis population. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). Confidence intervals (CI) were calculated using the exact (Clopper-Pearson) method.
Time Frame: Up to approximately 10 months
Population: Modified intent-to-treat (mITT) population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 7 | 6
Percentage of Participants | 0 [0 to 41] | 0 [0 to 45.9]

6. Secondary Outcome: Progression-free Survival (PFS) Per RECIST Version 1.1 by Investigator Assessment
Description: Progression free survival was defined as the interval between the date of T cell infusion and the earliest date of disease progression or death due to any cause. Progressive disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. PFS based on responses assessed by investigator per RECIST v1.1 is presented. Kaplan-Meier Median and 95% confidence intervals are presented. Confidence intervals were calculated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 10 months
Population: Modified intent-to-treat (mITT) population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 7 | 6
Months | 5.32 [1.45 to 5.52] | 1.48 [0.62 to 2.83]

7. Secondary Outcome: Disease Control Rate (DCR) Per RECIST Version 1.1 by Investigator Assessment
Description: DCR was defined as the percentage of participants with a confirmed complete response (CR), partial response (PR), or stable disease (SD) for at least 6 months as per RECIST v1.1. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Confidence intervals (CI) were calculated using the exact (Clopper-Pearson) method.
Time Frame: Up to approximately 10 months
Population: Modified intent-to-treat (mITT) population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 7 | 6
Percentage of Participants | 0 [0 to 41] | 0 [0 to 45.9]

8. Secondary Outcome: Duration of Response (DOR) Per RECIST Version 1.1 by Investigator Assessment
Description: Duration of response was defined as the interval between the initial date of confirmed response (PR/CR) and the date of progressive disease or death among participants with a confirmed response per RECIST 1.1. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters.
Time Frame: Up to approximately 10 months
Population: Modified intent-to-treat (mITT) population. Only participants with CR or PR were included in the analysis. No participant achieved CR or PR, hence the number of participants analyzed is 0.
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Response (TTR) Per RECIST Version 1.1 by Investigator Assessment
Description: Time to response was defined as the interval of time between the date of T-cell infusion and the first documented evidence of the confirmed response (PR or CR), in the subset of participants with a confirmed PR or CR as their best confirmed overall response. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm.
Time Frame: Up to approximately 10 months
Population: as for outcome 8
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Maximum Transgene Expansion (Cmax) of Lete-cel
Description: Cmax was defined as peak cell expansion during the study. Blood samples were collected for analysis of Cmax of lete-cel.
Time Frame: Day 1 to Day 15
Population: Pharmacokinetic (PK) population included all participants in the mITT population from whom at least one PK sample was obtained, analyzed, and was measurable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies per microgram genomic DNA
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 7 | 6
Copies per microgram genomic DNA | 155712.1398 (55.21519) | 127343.0679 (34.95574)

11. Secondary Outcome: Time to Cmax (Tmax) of Lete-cel
Description: Tmax was defined as time to reach peak cell expansion during the study. Blood samples were collected for analysis of Tmax of lete-cel.
Time Frame: Day 1 to Day 15
Population: Pharmacokinetic (PK) population
Measure: Median (Full Range); unit: Days
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 7 | 6
Days | 3 [1 to 15] | 7.9 [1 to 15]

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve to Day 28 (AUC0-28d) of Lete-cel
Description: Area under the cell expansion-time curve from first T-cell infusion to Day 28. Blood samples were collected to measure AUC (0-28 days).
Time Frame: Up to 28 days
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*copies per microgram genomic DNA
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab
Number analyzed (Participants) | 7 | 6
Days*copies per microgram genomic DNA | 1646416.5835 (109.45757) | 1565617.646 (46.16918)

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to approximately 10 months
Description: All cause mortality , SAEs and non-serious adverse events were reported for the Intent to Treat (ITT) population that includes all participants who started the leukapheresis procedure. Participants in the "No Treatment" arm started the leukapheresis procedure but did not receive lymphodepletion chemotherapy or Lete-cel infusion.
Groups:
- No Treatment: Participants who underwent leukapheresis but did not go on to receive lymphodepletion chemotherapy or T-cell infusion.
Arm/Group | Arm A: Lete-cel Monotherapy | Arm C: Lete-cel + Pembrolizumab | No Treatment
All-Cause Mortality (participants affected / at risk) | 3/7 | 1/6 | 5/21
Serious Adverse Events (participants affected / at risk) | 5/7 | 4/6 | 2/21
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 3/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Lete-cel Monotherapy (N=7) | Arm C: Lete-cel + Pembrolizumab (N=6) | No Treatment (N=21)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Lete-cel Monotherapy (N=7) | Arm C: Lete-cel + Pembrolizumab (N=6) | No Treatment (N=21)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 5 (5) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 4 (4) | 4 (5) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (6) | 0 (0) | 0 (0)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood fibrinogen increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood methaemoglobin present (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (8) | 4 (4) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (4) | 4 (4) | 0 (0)
Platelet count decreased (Investigations) | 4 (5) | 1 (1) | 0 (0)
Serum ferritin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (3) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 6 (7) | 2 (3) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 3 (3) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (4) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (12) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (3) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT03709706/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT03709706/SAP_001.pdf